CLINICAL TRIAL: NCT03553641
Title: The Effect of Dental Hyperalgesia and Mechanical Allodynia on Assessment Capacity of Patients in a Local Turkish Population
Brief Title: The Effect of Central Sensitization on Assessment Capacity of Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Tan Firat Eyuboglu, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: 404
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Symptomatic Irreversible Pulpitis; Acute Apical Periodontitis of Pulpal Origin
Keywords: capacity; clinical ethics; autonomy; competence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of this study is to evaluate the effect of dental hyperalgesia and mechanical allodynia on the assessment capacity of individuals in a local Turkish population. The hypothesis of this study is that excessive amounts of pain and a major functional shift in the somatosensory system due to central sensitization might cause unwitting intent.

DETAILED DESCRIPTION:
It included patients between the ages of 18 and 70 who had a symptomatic tooth in need of non-surgical root canal treatment. All enrolled subjects volunteered and signed a written informed consent. Patients diagnosed with systemic diseases and those who had used an analgesic within 12 hours prior to the appointment were excluded from the study. A total of 30 patients were included in the study. A data sheet including patients' demographic data, diagnostic data, and data of explicit declaration of intent was completed. All pain scores were recorded according to the Visual Analog Scale (VAS). After the demographic data, diagnostic data. Patients were explicitly informed that the answers they were going to provide to the questions related to their explicit declaration of intent would not affect their diagnosis or the treatment they would undergo.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 18 and 70 who had a symptomatic tooth in need of non-surgical root canal treatment. All enrolled subjects volunteered and signed a written informed consent

Exclusion Criteria:

* Patients diagnosed with systemic diseases and those who had used an analgesic within 12 hours prior to the appointment were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: non
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
pain explicit declaration of intent | 30 minutes
  presence or absence of dental hyperalgesia and mechanical allodynia was recorded as well as the intensity of pain according to visual analog scale (VAS) with patients request of treatment to further evaluate any relevance between the variables. VAS scale is between 1 to 10 and 1 means no pain and 10 means worst pain ever. The scale was drawn as a 10 cm line on a paper, with a number at the beginning of each cm from 1 to 10 and patients were asked to show the respected place regarding their intensity of pain they were experiencing on the line.

SECONDARY OUTCOMES:
aesthetics | 30 minutes
  patient who chose extraction were asked their choice of treatment if the relevant tooth were to be an anterior tooth and recorded as yes or no
previous RCT | 30 minutes
  patients were asked if they had any root canal treatment previously and recorded as yes or no
excessive pain | 30 minutes
  patient who chose extraction were asked their choice of treatment if the painh were not to be excessive and recorded as yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Tan F EYUBOGLU, PROF, Principal Investigator — Istanbul Medipol University Faculty of Dentistry; Fulya I GONENC, PROF, Principal Investigator — Istanbul Medipol University Faculty of Law
Locations (1):
- İstanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
name of the study and name of the researchers

REFERENCES:
- [Background] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153